CLINICAL TRIAL: NCT06852547
Title: Ingestion of a Novel Algae Protein Source on Rested and Post Exercise Muscle Protein Synthesis Rates.
Brief Title: The Effect of Ingesting a Novel Algae Protein Source on Rested and Exercised Muscle Protein Synthesis Rates in Older Adults.
Acronym: CALM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Principal Investigator, Freyja Haigh, Postdoctoral Research Associate, University of Exeter
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 9071916
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Nutritional Intervention
Keywords: novel protein; protein synthesis; older adults; alge
MeSH Terms: interventions — Proteins; 95-kDa protein, green algae

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Whey protein (Active Comparator)
  Interventions: Dietary Supplement: protein
- Algae protein (Experimental)
  Interventions: Dietary Supplement: protein

INTERVENTIONS:
Dietary Supplement: protein — protein
  Other Names: algae protein

SUMMARY:
To assess the rested and postexercise muscle protein synthetic response following the ingestion of a flavourless algae protein source compared with whey protein in older adults.

ELIGIBILITY:
Inclusion Criteria:

Males and Females BMI 18.5 - 30 kg/m2 Aged 65-80 years Recreationally Active

Exclusion Criteria:

Body mass index (BMI) <18.5 or >30 kg/m2 Any metabolic impairments Any cardiovascular impairments High blood pressure (≥140/90 mmHg) Any gastrointestinal disorders Any medications known to affect protein and/or amino acid metabolism A personal or family history of epilepsy, seizures or schizophrenia, motor disorder Chronic over the counter use of pharmaceuticals (> 1 month) Allergic to any of the whole foods included in the study

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-02-23 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Postprandial muscle protein synthesis | 4 hours
  unilateral exercise followed by protein ingestion (algae / whey)

CONTACTS AND LOCATIONS:
Locations (1):
- Health and Life Sciences, Exeter, United Kingdom

IPD SHARING:
Plan to Share IPD: No